CLINICAL TRIAL: NCT02395068
Title: Pharmacokinetics Study of Nimotuzumab Single-dose and Multiple-dose in Combination With Irinotecan in Patients With Solid Tumors
Brief Title: Pharmacokinetics Study of Nimotuzumab in Patients With Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Biotech Pharmaceutical Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BT-PK-001
Record Dates: First submitted 2015-02-28; First posted 2015-03-20 (Estimated); Last update posted 2015-08-19 (Estimated); Status verified 2012-10

CONDITIONS: Solid Tumors
Keywords: Pharmacokinetics; Nimotuzumab; Safety; Effcacy; Irinotecan
MeSH Terms: interventions — nimotuzumab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Single-dose PK (Experimental): single dose of nimotuzumab (100、200、400、600mg), with 3 weeks observation. 1 week after nimotuzumb administration, irinotecan (CPT-11) will be given at a dose of 180 mg/m2 once every 2 weeks, 2 weeks a cycle.
  Interventions: Drug: Nimotuzumab; Drug: irinotecan
- Weekly fixed dose (Experimental): Set 4 dose groups for Nimotuzumab, namely 100,200,400,600mg. Each group administered once a week for 6 weeks.
  Interventions: Drug: Nimotuzumab
- Bioweekly fixed dose PK (Experimental): Nimotuzumab 600mg, administered once every 2 weeks for 8 weeks. Dosing regimens can be adjusted according to the results of preliminary experiments. Nimotuzumab combined with irinotecan (180mg/m2), administering once every 2 weeks and considering 2 weeks as a period. If chemotherapy and Nimotuzumab are administered in the same day, chemotherapy should be infused after Nimotuzumab for at least 1h
  Interventions: Drug: Nimotuzumab; Drug: irinotecan

INTERVENTIONS:
Drug: Nimotuzumab — single dose of nimotuzumab (100、200、400、600mg), with 3 weeks observation；Set 4 dose groups for Nimotuzumab, namely 100,200,400,600mg. Each group administered once a week for 6 weeks；600mg, administered once every 2 weeks for 8 weeks.
  Other Names: Taixinsheng
Drug: irinotecan — Single-dose PK：1 week after nimotuzumb administration, irinotecan (CPT-11) will be given at a dose of 180 mg/m2 once every 2 weeks, 2 weeks a cycle.
  Bioweekly fixed dose PK：Nimotuzumab combined with irinotecan (180mg/m2), administering once every 2 weeks and considering 2 weeks as a period. If chemotherapy and Nimotuzumab are administered in the same day, chemotherapy should be infused after Nimotuzumab for at least 1h
  Other Names: CPT-11
  Arms: Bioweekly fixed dose PK; Single-dose PK

SUMMARY:
Nimotuzumab is an IgG1 humanized monoclonal antibody that recognized an epitope located in the extra cellular domain of the human epidermal growth factor receptor (EGFR), inhibiting tyrosine kinase activation. It has been approved to treat squamous cell carcinoma of head and neck (SCCHN), glioma and nasopharyngeal carcinoma in different countries. Currently, the registered clinical trials of Nimotuzumab combined with chemotherapy in advanced non-small cell lung cancer, colorectal cancer, esophageal cancer and glioma have been approved and are ongoing all over the investigators' country. The main purpose of this study is to evaluate the pharmacokinetic characteristics of Nimotuzumab combined with Irinotecan in patients with solid tumors.

DETAILED DESCRIPTION:
This is a single-centered, non-randomized and open-labeled Clinical Pharmacokinetics Study of Nimotuzumab in patients with solid tumors. The test includes 3 dose groups, namely Single dose group, Multiple single-week dose group and Multiple bi week dose group, to evaluate the pharmacokinetic characteristics of Nimotuzumab combined with Irinotecan in patients with solid tumors.

ELIGIBILITY:
Inclusion criteria:

1. Confirmed by pathology and / or cytology diagnosis in patients with advanced solid tumors
2. Failure of first-line or multi-line chemotherapy and be suitable for irinotecan therapy
3. Age 18-70 years, both genders at enrollment
4. ECOG 0 to 1
5. Adequate bone marrow function
6. Recover from the toxicity of previous treatment
7. At least one measurable site of disease as defined by at least 20mm in greatest dimension by CT or 10mm in greatest dimension by SCT/MRI
8. Male or female with fertility in the trial are willing to take contraceptive measures
9. Estimated life expectancy of 3 months or greater
10. All patients signed written informed consent

Exclusion criteria:

1. Have previously received EGFR-targeted therapy
2. Current treatment on other effective programs
3. Participated in other clinical trial within 4 weeks after enrollment
4. Nervous system symptoms caused by brain metastases need to apply steroidal anti-edema medications to control
5. Persistent uncontrollable diarrhea CTCAE 2 level and above (4-6 times daily)
6. Complete or incomplete intestinal obstruction
7. Need to drainage pleural effusion and ascites
8. Drug addiction and other adverse long-term alcoholics, as well as AIDS patients
9. Occurred myocardial infarction within 6 months
10. Diagnosed with severe interstitial pneumonitis or pulmonary fibrosis by Chest CT
11. Severe or uncontrolled complications, such as infection required systemic treatment，fever（≥38℃），congestive heart failure，diabetes or hypertension that can not be controlled by drugs and other complications that may interfere with drug efficacy
12. Drug allergy（≥CTCAE 3.0）, such as shock or allergy symptoms, especially allergic to similar drugs in the past and severe hypersensitivity to polysorbate eighty-containing drugs
13. Uncontrollable seizures or loss of insight because of psychosis
14. Female patient is pregnant, breastfeeding, or of childbearing potential but not take contraceptive measures
15. Male patient who want his spouse to be pregnant during the trial
16. Researchers believe that should not participate in this trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-11 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics of Nimotuzumab after administration of escalating single dosing and weekly fixed dosing in patients with solid tumors: Single dose：Tmax，Cmax， AUC，Vc，t1/2α，t1/2β，CL. Multiple dose：Tmax，Css-min，Css-max，Css-a，t1/2β，CL，AUCss，DF. | up to 9 weeks
  The measure is a composite.The measure of single dose：Tmax，Cmax， AUC，Vc，t1/2α，t1/2β，CL.
  The measure of multiple dose：Tmax，Css-min，Css-max，Css-a，t1/2β，CL，AUCss，DF.

SECONDARY OUTCOMES:
Safety - AE measured by NCI CTCAE v 3.0 | Any adverse medical events occur from the beginning of receiving study drug to the end of treatment after 30 days
  Safety evaluations included adverse events and changes in laboratory data.Adverse events were descriptive statistics, lists the event occurred, the duration, severity, and drug relationship, as well as its outcome.
ORR（Objective Response Rate） | The third weekend and Ninth weekend
  Efficacy as measured by RECIST v1.1
DCR（Disease Control Rate） | The third weekend and Ninth weekend
  Efficacy as measured by RECIST v1.1
PFS（Progression Free Survival） | The third weekend and Ninth weekend
  Efficacy as measured by RECIST v1.1

CONTACTS AND LOCATIONS:
Overall Officials: Jinwan Wang, PhD，MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Cancer Institute & Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China